CLINICAL TRIAL: NCT01993849
Title: A Randomized Placebo-controlled Trial of N-Acetylcysteine in Onychophagia
Brief Title: Use of N-Acetylcysteine (NAC) in Fingernail Biting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kevin Gray, MD (Other)
Responsible Party: Sponsor-Investigator, Kevin Gray, MD, Associate Professor, Medical University of South Carolina
Organization: Medical University of South Carolina (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00028506
Record Dates: First submitted 2013-09-24; First posted 2013-11-25 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Onychophagia
Keywords: Anxiety; Impulse control; Depression; ADHD; Fingernail Biting; N-Acetylcysteine; NAC
MeSH Terms: conditions — Nail Biting; Anxiety Disorders; Depression; Attention Deficit Disorder with Hyperactivity | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- N-Acetylcysteine (NAC) (Active Comparator): Oral N-acetylcysteine 1200 mg twice daily dosing for 8 weeks
  Interventions: Drug: N-Acetylcysteine (NAC)
- Placebo (Placebo Comparator): Oral placebo (matched in appearance to active treatment) twice daily dosing for 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: N-Acetylcysteine (NAC) — This is the medication N-acetylcysteine (NAC)
  Other Names: NAC
  Arms: N-Acetylcysteine (NAC)
Other: Placebo — Placebo, designed to match in appearance to NAC
  Arms: Placebo

SUMMARY:
To conduct a pilot randomized placebo-controlled feasibility trial of N-acetylcysteine (NAC) in onychophagia, preliminarily assessing the tolerability and effects of this pharmacotherapy on young adults who bite their fingernails. It is proposed that NAC will help decrease fingernail biting.

DETAILED DESCRIPTION:
This is a proof-of-concept pilot placebo-controlled trial of N-acetylcysteine (NAC) in young people who bite fingernails. The primary interest is in assessing the feasibility of conducting this line of research, while preliminarily exploring potential effects on nail biting, as measured by nail length.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-30 2. Fingernail biter for ≥5 years

Exclusion Criteria:

* 1. Any unstable major DSM-IV Axis I psychiatric disorder in the past month (e.g., psychotic disorders, bipolar disorder, major depressive disorder) 2. Current substance dependence in the past month 3. Current unstable major medical disorder or medical condition in the past 6 months (e.g., renal impairment) 4. Current pregnancy or breastfeeding 5. Current seizure disorder or asthma, due to possible elevated risk for adverse effects with NAC in individuals with these conditions 6. Known hypersensitivity to NAC 7. Use of carbamazepine or nitroglycerin (or any other medication deemed to be hazardous if taken with NAC) within 14 days of study participation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Gray, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- N-Acetylcysteine: Twice daily dosing for 8 weeks
  N-Acetylcysteine (NAC)
- Placebo: Twice daily dosing for 8 weeks
  Placebo
Period: Overall Study
Arm/Group | N-Acetylcysteine | Placebo
Started | 12 | 11
Completed | 9 | 9
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- N-Acetylcysteine (NAC): 1200 mg twice daily dosing for 8 weeks
  N-Acetylcysteine (NAC)
- Total: Total of all reporting groups
Arm/Group | N-Acetylcysteine (NAC) | Placebo | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (5.2) | 27.4 (4.7) | 27.0 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Enrolled Within One Year
Description: Ability to enroll the goal sample within one year; we are interested in the feasibility of sufficient enrollment and data collection within a given period of time.
Time Frame: 1 year
Population: The goal sample was to enroll at least 10 participants per arm/group within the specified recruitment period.
Measure: Count of Participants; unit: Participants
Arm/Group | N-Acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 12 | 11
Participants | 12 | 11

2. Other Pre Specified Outcome: Measurement of Nail Length
Description: Length of nails, measured by caliper
Time Frame: End of 8-week treatment
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- N-Acetylcysteine: 1200 mg twice daily dosing for 8 weeks
  N-Acetylcysteine (NAC)
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 12 | 11
millimeters | 10.12 (2.43) | 10.73 (3.40)
Statistical Analysis 1: Comparison: N-Acetylcysteine vs Placebo; Test type: Superiority; p = 0.69, t-test, 2 sided — The p-value was calculated, and is not attempting to indicate the threshold for statistical significance; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [-3.81 to 2.59]

ADVERSE EVENTS:
Arm/Group | N-Acetylcysteine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 1/12 | 0/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetylcysteine (N=12) | Placebo (N=11)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No